CLINICAL TRIAL: NCT00996905
Title: Does Ultrasound Scanning of the Lumbar Spine Improve Patient Satisfaction and the Ease of Insertion of Labour Epidural Catheters
Brief Title: Does Ultrasound Scanning of the Lumbar Spine Improve Patient Satisfaction and the Ease of Insertion Epidurals?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Dr. Jose Carvalho, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-02
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Labor Pain
Keywords: Epidural Analgesia; Ultrasound; Training, Inservice
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Beginner Conventional (BC) (No Intervention): Beginner level (residents) doing epidural insertions the conventional way (ie. no ultrasound scanning)
- Beginner Ultrasound (BU) (Experimental): Beginner level (residents) doing epidural insertions with the help of ultrasound scanning.
  Interventions: Device: Portable ultrasound machine
- Experienced Conventional (No Intervention): Experienced level (fellows) doing epidural insertions the conventional way.
- Experienced Ultrasound (Experimental): Experienced level (fellows) doing epidural insertions with the help of ultrasound scanning.
  Interventions: Device: Portable ultrasound machine

INTERVENTIONS:
Device: Portable ultrasound machine — Each patient will have their lumbar spine scanned by ultrasound for a maximum period of 5 minutes.
  Arms: Beginner Ultrasound (BU)
Device: Portable ultrasound machine — Each patient will have their lumbar spine scanned by ultrasound for a maximum period of 5 minutes.
  Arms: Experienced Ultrasound

SUMMARY:
Ultrasound scanning of the back has been shown to increase success when used to guide epidural catheter insertion. However, this technique is not applied widely in clinical practice. Stronger evidence is required to prove that it will improve the clinical experience of labour epidurals.

The study hypothesis is that anesthesiologists (both residents and fellows), will have an increased rate of success and ease of insertion of labour epidural catheters, and that there will be increased patient satisfaction, if ultrasound scanning of the lumbar spine is done prior to the procedure.

DETAILED DESCRIPTION:
Studies have shown that ultrasound scanning of the lumbar spine is beneficial in certain circumstances (eg. predicted difficult epidurals). However, no large scale studies with multiple anesthesiologists performing the technique have been done to show that ultrasound scanning may be of benefit in their everyday clinical practice.

This study will involve residents and fellows, each performing epidural insertions with and without the use of ultrasound scanning of the lumbar spine prior to the procedure. If the hypothesis is correct, then the use of this technique may become widespread, resulting in less complications and increased patients satisfaction.

ELIGIBILITY:
For Patients:

Inclusion Criteria:

* ability to Speak in English
* requesting epidural analgesia for labour
* having easily palpable spine (clinically 'easy' back)

Exclusion Criteria:

* contraindications to epidural analgesia
* patients with a history of difficult epidural insertions or spinal anesthetic
* Patients with a known history of back surgery
* patients with known significant kyph0scoliosis

For Anesthesiologists:

Inclusion Criteria:

* Residents and fellows training or practicing at Mount Sinai hospital and enrolled in either a residency or fellowship program at the University of Toronto.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Ease of epidural insertion by the following 3 measurements: time to perform procedure (minutes), number of levels at which insertion is attempted, and number of ventral passes of the epidural needle. | 20 minutes

SECONDARY OUTCOMES:
The occurrence of inadvertent dural punctures. | 24-48 hours
Number of attempts to thread the epidural catheter | 20 minutes
Success or failure of the epidural (defined as lack of sufficient analgesia within 2 hours of insertion, necessitating re-insertion) | 2 hours
The need of the anesthesiologist to call for assistance with the procedure | 30 minutes
Patient satisfaction as determine by a questionnaire | 24 hours and 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Arzola C, Mikhael R, Margarido C, Carvalho JC. Spinal ultrasound versus palpation for epidural catheter insertion in labour: A randomised controlled trial. Eur J Anaesthesiol. 2015 Jul;32(7):499-505. doi: 10.1097/EJA.0000000000000119. PMID 25036283